CLINICAL TRIAL: NCT00510120
Title: Mediators, Moderators, and Treatment Outcomes With ODD Youth
Brief Title: Comparison of Two Psychosocial Therapies for Treating Children With Oppositional-Defiant Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas H. Ollendick, University Distinguished Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH076141 (NIH); R01MH076141 (NIH); DDTR B3-PDC
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Oppositional-Defiant Disorder
Keywords: Attention Deficit and Disruptive Behavior Disorders; Conduct Disorder; Behavior Problems in Youth; Argumentativeness; Children; Therapy; Attention Deficit Disorder
MeSH Terms: conditions — Oppositional Defiant Disorder; Attention Deficit and Disruptive Behavior Disorders; Conduct Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive collaborative problem solving.
  Interventions: Behavioral: Collaborative problem solving (CPS)
- 2 (Active Comparator): Participants will receive parent management training.
  Interventions: Behavioral: Parent management training (PMT)
- 3 (Active Comparator): Participants assigned to waitlist control will receive one of the two treatments after a 10-weeks waitlist period.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Parent management training (PMT) — PMT primarily involves teaching parents strategies to respond consistently and correctly to their child's behavior. Parents assigned to the PMT group will be taught how to respond consistently and appropriately to their child's positive and negative behaviors. Participants will attend a 1-hour treatment session each week for 10 weeks.
  Other Names: PMT
  Arms: 2
Behavioral: Collaborative problem solving (CPS) — CPS is a treatment approach that involves both the parent and child by teaching parents to help their child control their emotions and to problem solve as a family. Parents assigned to the CPS group will be taught strategies to help their child identify and regulate emotions and to solve behavior problems together as a family. Participants will attend a 1-hour treatment session each week for 10 weeks.
  Other Names: CPS
  Arms: 1
Behavioral: Waitlist control — Participants assigned to the waitlist control condition group will wait 10 weeks before beginning treatment one of the two treatment options.
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness of two different psychosocial therapies, parent management training and collaborative problem solving, in treating children with oppositional-defiant disorder.

DETAILED DESCRIPTION:
Oppositional-defiant disorder (ODD) is characterized by a recurrent pattern of developmentally inappropriate levels of negative, defiant, disobedient, and hostile behavior toward authority figures. Behaviors associated with ODD include temper tantrums; persistent stubbornness; resistance to directions; unwillingness to compromise, give in, or negotiate; deliberate or persistent testing of limits; and verbal and minor physical aggression. The usual treatment approach for children with ODD is parent management training (PMT). PMT primarily involves teaching parents strategies to respond consistently and correctly to their child's behavior. However, PMT does not always lead to longstanding results and there is a need for alternative treatments. Collaborative problem-solving (CPS) is a treatment approach that involves both the parent and child by teaching parents to help their child control their emotions and to problem-solve as a family. This study will compare the effectiveness of CPS and PMT in treating children with ODD.

Participants in this open-label study will include children with ODD and their parents. Participants will be randomly assigned to one of three groups: CPS, PMT, or waitlist control. Parents assigned to the CPS group will be taught strategies to help their child identify and regulate emotions and to solve behavior problems together as a family. Parents assigned to the PMT group will be taught how to respond consistently and appropriately to their child's positive and negative behaviors. Participants assigned to the waitlist control condition group will wait 10 weeks before treatment begins. Participants will attend a 1-hour treatment session each week for 10 weeks. In order to determine whether treatment is effective, participants will be asked to complete a variety of questionnaires, talk with their child about solving problems, and complete a structure diagnostic interview prior to the beginning of treatment, following treatment, and at a 1-year follow-up session. Parents will be asked to submit their child's school grades and school attendance records. If granted permission by the parents, the child's teacher will complete a questionnaire regarding the child's behavior in school for the year prior to participating in the study and up to 1 year after treatment. The information collected will help to determine how treatment affects each child's progress.

ELIGIBILITY:
Inclusion Criteria for Children:

* Meets DSM-IV criteria for oppositional-defiant disorder
* Parent or guardian willing to provide informed consent

Exclusion Criteria for Children:

* History or current diagnosis of CD, autism, pervasive developmental disorders (PDD), or any psychotic disorder
* An estimated Full Scale IQ below 80
* Current suicidal or homicidal ideation

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2007-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
ODD, conduct disorder (CD), and attention deficit hyperactivity disorder (ADHD) using a Diagnostic Interview Schedule for Children | Measured at Year 1 follow-up visit
Disruptive Behavior Disorders Rating Scale | Measured at Year 1 follow-up visit

SECONDARY OUTCOMES:
Behavior Assessment System for Children | Measured at Year 1 follow-up visit
Parent Satisfaction Questionnaire: Parental satisfaction with the treatment approach and the strategies they use to discipline their children in terms of both difficulty and usefulness | Measured at Weeks 4 and 7, immediately post-treatment, and Year 1 follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H. Ollendick, PhD, Principal Investigator — Department of Psychology, Virginia Tech
Locations (1):
- Child Study Center, Blacksburg, Virginia, United States